CLINICAL TRIAL: NCT03351400
Title: Japanese OMI Treatment With Kit-positive Cells for Enhanced Regeneration Trial
Brief Title: Japanese OMI Treatment With Kit-positive Cells for Enhanced Regeneration
Acronym: JOKER
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sakakibara Heart Institute (Other)
Collaborators: CellBank of Japan (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB3170012
Record Dates: First submitted 2017-11-14; First posted 2017-11-22 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Chronic Heart Failure; Old Myocardial Infarction
Keywords: cardiac stem cells; c-kit
MeSH Terms: conditions — Piebaldism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Stem cells administered to participants
  Interventions: Biological: Stem cells administered to participants

INTERVENTIONS:
Biological: Stem cells administered to participants — Patients in this arm will receive intracoronary infusion of 1,000,000 autologous c-kit positive cardiac stem cells.

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of intracoronary infusion of autologous cardiac stem cells in patients with ischemic cardiomyopathy.

DETAILED DESCRIPTION:
This phase I trial will involve 6 patients suffering from chronic ischemic cardiomyopathy and congestive heart failure, to be compared with historical control subjects. This study will be conducted as a collaborative project between the Sakakibara Heart Institute and the CellBank of Japan. The trial is designed to assess the safety and effectiveness of autologous administration of 1,000,000 c-kit-positive cardiac stem cells (CSCs) via intracoronary route following cultivation. The preliminary eligibility criteria will utilize a left ventricular ejection fraction (LVEF) less than 40% measured by echocardiography. During the coronary artery bypass grafting (CABG) surgery, a part (less than 1 gram) of the right atrial appendage (RAA) will be harvested and frozen. When the LVEF is less than 40% after the CABG surgery, the subject will be enrolled as a candidate for the delivery of CSCs, which will be selected from the RAA tissue and cultured for a few months for expansion. The outcome will be evaluated by adverse events as well as cardiac functions.

ELIGIBILITY:
Inclusion Criteria:

* Adult with ability to provide informed consent.
* Left ventricular ejection fraction less than 40% as evidenced by echocardiogram.
* Scheduled for elective surgical revascularization within 2 months.

Exclusion Criteria:

* Positive for HBs-Ag, HCV-Ab, HIV-Ab, or tests for syphilis.
* Diabetic HbA1c greater than 8.5%.
* Pregnant women.
* Scheduled for additional interventions including ventriculoplasty.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2017-11-15 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Monitoring adverse events | 2 years
  Including death, ventricular arrhythmia, bleeding, myocardial infarction, cardiac tumor, brain stroke, peripheral embolism

SECONDARY OUTCOMES:
NYHA classification | 2 years
  Measurement of symptom
Serum NT-proBNP | 2 years
  Measurement of cardiac function
Electrocardiogram | 2 years
  Measurement of arrhythmia
Chest X-ray | 2 years
  Measurement of cardiac function
Cardiopulmonary exercise test | 2 years
  Measurement of cardiopulmonary function
Echocardiogram | 2 years
  Measurement of cardiac function
Magnetic resonance imaging | 2 years
  Measurement of cardiac function
Myocardial scintigraphy | 2 years
  Measurement of myocardial viability

CONTACTS AND LOCATIONS:
Locations (1):
- Sakakibara Heart Institute, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chugh AR, Beache GM, Loughran JH, Mewton N, Elmore JB, Kajstura J, Pappas P, Tatooles A, Stoddard MF, Lima JA, Slaughter MS, Anversa P, Bolli R. Administration of cardiac stem cells in patients with ischemic cardiomyopathy: the SCIPIO trial: surgical aspects and interim analysis of myocardial function and viability by magnetic resonance. Circulation. 2012 Sep 11;126(11 Suppl 1):S54-64. doi: 10.1161/CIRCULATIONAHA.112.092627. PMID 22965994